CLINICAL TRIAL: NCT06174649
Title: Fast Antibiotic Susceptibility Testing for Gram Negative Bacteremia Trial
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Parexel (Industry); BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Pro00109586; UM1AI104681 (NIH)
Record Dates: First submitted 2023-12-05; First posted 2023-12-18 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2024-12

CONDITIONS: Gram-negative Bacteremia; Bloodstream Infection
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Patient and care provider will not know which arm subject is randomized into until after the stewardship team has review the Reveal results and provided feedback on initial therapies prescribed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): When a blood culture growing GNB is randomized standard of care arm the positive blood cultures will be characterized using standard of care antimicrobial susceptibility testing (AST)
- Reveal (Active Comparator): When a blood culture growing GNB is randomized to the Reveal arm, the positive blood culture will be characterized using Reveal, a rapid AST, and the standard of care AST.
  Interventions: Diagnostic Test: Reveal

INTERVENTIONS:
Diagnostic Test: Reveal — Reveal is a rapid AST method, which uses small molecule sensor technology to detect growth of bacterial populations by measuring volatile metabolites, and provides AST results in ~5 hours. Reveal™ is approved for clinical use in the European Union (EU) and Israel and approval is in process in India, and provides minimum inhibitory concentrations (MICs) for 28 antibiotics and 9 Gram negative species, that together account for ~90% of organisms causing Gram negative blood stream infections (BSI).
  Arms: Reveal

SUMMARY:
This study is a 2-arm, multicenter, multinational, prospective, randomized, controlled clinical trial. Hospitalized subjects with blood cultures growing Gram negative bacilli (GNB) will be randomized 1:1 to have the positive blood cultures characterized using standard of care (SOC) antimicrobial susceptibility testing (AST) vs. a rapid AST method known as Reveal™ in addition to SOC AST. The purpose of the FAST trial is to evaluate whether use of a rapid phenotypic AST improves clinical outcomes compared to use of SOC AST methods in clinical settings with high resistance rates.

ELIGIBILITY:
Inclusion Criteria:

1. Positive blood culture with Gram stain showing GNB
2. Hospitalized at the time of Gram stain result
3. Enrolled within 16 hours of blood culture positivity

Exclusion Criteria:

1. Positive blood culture for GNB within the prior 7 days (if known at the time of Gram stain result)
2. Deceased at the time of Gram stain result
3. Gram-positive bacilli, Gram-positive cocci, Gram-negative cocci, yeast, fungi, or multiple morphologies of GNB detected on Gram stain of blood culture
4. Previous enrollment in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2023-12-22 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Subject Clinical Outcomes, as measured by Desirability of Outcome Ranking (DOOR) | Up to 30 days after Gram stain result
  The composite 3-category DOOR outcome will assess three deleterious events (unsuccessful discharge, lack of clinical response, and undesirable events) in addition to survival up to 30 days after Gram stain result. The primary DOOR outcome measure is defined using three ordered levels. From best to worst, they are:
  1. Alive without deleterious events
  2. Alive with at least 1 deleterious event
  3. Death

SECONDARY OUTCOMES:
All-Cause Mortality | Up to 30 days post Gram Stain
  All-cause in-hospital mortality up to 30 days post Gram stain result
Hospital Stay Length | up to 30 days post Gram stain result
  Length of index stay in the hospital up to 30 days post Gram stain result, for those subjects alive at 30 days. Length of stay will be calculated as date of discharge minus date of Gram stain result.
Number of ICU admissions | up to 30 days post Gram stain result
  ICU admission up to 30 days post Gram stain result
Number of participants with new Acquisition of Multi-Drug Resistant Organism (MDRO) and/or C. difficile | up to 30 days post Gram stain result
  New acquisition is defined as detection of MDRO/C. difficile in subjects who do not have preceding clinical or surveillance cultures with these organisms in the prior 3 months. MDRO will be identified on routine clinical or surveillance samples using local laboratory diagnostic procedures and include:
  Methicillin-resistant Staphylococcus aureus Vancomycin-resistant Enterococcus species 3rd generation cephalosporin-non-susceptible Enterobacterales Carbapenem-resistant Enterobacterales, as defined by the Center for Disease Control and Prevention: resistant to imipenem, meropenem, doripenem, or ertapenem OR documentation that the isolate produces a carbapenemase Pseudomonas aeruginosa resistant to carbapenems/multi-drug resistant (resistant to aminoglycosides, cephalosporins, fluoroquinolones, and carbapenems) Carbapenem-resistant Acinetobacter species Candida auris
Time to effective antibiotic therapy | within 3 days from Gram stain result
  Time to effective antibiotic therapy within 3 days from Gram stain result, defined as treatment with an antibiotic (or antibiotic class) to which the blood isolate is susceptible based on standard of care (SOC) AST.
Time to antibiotic escalation | within 3 days from Gram stain result
  Time to antibiotic escalation of Gram negative coverage in those who have antibiotic escalation within 3 days from Gram stain result.
  Escalation: Changing to a broader spectrum antibiotic, addition of one or more antibiotics, or conversion of oral (PO) to intravenous (IV) route.
Time to antibiotic de-escalation of Gram negative coverage | within 3 days from Gram stain result
  Time to antibiotic de-escalation of Gram negative coverage in those who have antibiotic de-escalation within 3 days from Gram stain result.
  De-escalation: Changing to a narrower spectrum antibiotic , cessation of one or more antibiotics, or changing from an IV to PO route of appropriate drug (i.e. IV to PO ciprofloxacin or levofloxacin).

CONTACTS AND LOCATIONS:
Overall Officials: Ritu Banerjee, MD, PhD, Principal Investigator — Vanderbilt University Medical Center; Vance Fowler, MD, Study Director — Duke Clinical Research Institute
Locations (7):
- Greece (2):
  - Attikon University General Hospital, Chaïdári, Attica
  - Tzaneio General Hospital, Piraeus
- Kasturba Medical College, Mangalore, Attavāra, Mangalore, India
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Meir Medical Center, Kfar Saba
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Complexo Hospitalario Universitario A Coruña (CHUAC) Sergas, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banerjee R, Komarow L, Li Y, Wu Q, Sanchez-Gonzalez L, Mau D, Abbenante E, Schwager N, Dodd A, Souli M, Geres HS, Doernberg S, Greenwood-Quaintance K, Evans SR, Chambers HF, Fowler VG Jr, Patel R; Antibacterial Resistance Leadership Group. Study protocol for a multicenter, multinational prospective randomized controlled trial comparing outcomes in subjects with Gram-negative bacteremia who have blood culture evaluation using Fast Antibiotic Susceptibility Testing vs. standard of care testing: the FAST trial. Trials. 2025 Nov 12;26(1):500. doi: 10.1186/s13063-025-09228-4. PMID 41225518

DOCUMENTS (1):
  • Informed Consent Form (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT06174649/ICF_000.pdf